CLINICAL TRIAL: NCT01883687
Title: Functional Nasal Surgery at the Time of Le Fort I Osteotomy: A Prospective, Single-blind, Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102-0546C
Record Dates: First submitted 2013-05-23; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-04

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Septoplasty (Experimental): patients will receive septoplasty together with Le Fort I osteotomy
  Interventions: Procedure: Septoplasty
- No septoplasty (No Intervention): patient will only receive Le Fort I osteotomy

INTERVENTIONS:
Procedure: Septoplasty
  Arms: Septoplasty

SUMMARY:
Objectives: The aims of this study are (1) to define the effectiveness of functional nasal surgery during Le Fort I osteotomy on nasal obstruction through objective as well as subjective evaluations, (2) to determine guideline for concomitant functional nasal surgery with Le Fort I osteotomy, and (3) to explore possible mechanisms by which functional nasal surgery may reduce nasal obstruction severity.

Design: A prospective, single-blnd, randomized trial. Setting: Chang Gung Craniofacial Center and Department of Otolaryngology (ENT). Patients: A total of 80 Taiwanese patients with unilateral cleft lip and palate and dentofacial deformity (age >16 for females, >18 for males; 40 in experimental and 40 in control groups) Interventions: In the experimental group, all patients will receive Le Fort I osteotomy and septoplasty. In the control group, all patients will receive Le Fort I osteotomy only.

Measurements: All patients will undergo history taking, clinical examination, radioallergosorbent (RAST) examination (before surgery), standard questionnaire and image examination before surgery, one week, 1, 3, 6, 12 and 24 months after surgery. To reduce radiation exposure, cone-beam CT will only be performed before surgery and one week, 12 and 24 months after surgery.

Data Analysis: Independent t and chi-squared tests, correlation coefficients and repeated measures analysis of variance (ANOVA) will be used. Statistical significance is assumed for a p value of less than 0.05.

Key Words: cleft lip palate, nasal septum deviation, Le Fort I osteotomy, septoplasty, effectiveness

ELIGIBILITY:
Inclusion Criteria:

1. Taiwanese adults with dentofacial deformities (DFD)
2. Have documented nasal obstruction and a hypertrophied inferior turbinate on the contralateral side of the septal deviation
3. Will undergo bimaxillary surgery including 1-piece Le Fort I osteotomy for DFD at the Craniofacial Center between 2012 and 2013

Exclusion Criteria:

1. Previous OGS or nasal surgery
2. Patients with nasal polyposis, rhinosinusitis or neoplasia
3. Patients with clefts or craniofacial anomaly
4. Patients with adenoid hypertrophy, nasal valve collapse, uncontrolled asthma or tobacco use
5. Noncompliance for test
6. Noncompliance to test schedule
7. Won't sign informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Changes in symptom severity and health-related quality of life in sinonasal conditions | before surgery and 24 months after surgery
  Sino-Nasal Outcome Test 22(SNOT-22) questionnaire will be used

SECONDARY OUTCOMES:
Changes in nasal patency and congestion | before surgery and 24 months after surgery
  Acoustic rhinometry will be used
Changes of nasal airway volume | before surgery and 24 months after surgery
Changes in transnasal pressure and airway resistance and pressure-flow characteristics | before surgery and 24 months after surgery
  Rhinomanometry will be used
Changes of causative allergens | before surgery and 24 months after surgery
  RAST examination will be used

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Fang Liao, PHD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan